CLINICAL TRIAL: NCT06244745
Title: Clinical and Endocrinological Effects of Letrozole During the Luteal Phase After Controlled Ovarian Stimulation in Oocyte Donors: a Low Interventional, Randomized, Controlled Trial
Brief Title: Effects of Letrozole During the Luteal Phase After Controlled Ovarian Stimulation in Oocyte Donors.
Acronym: LETRODON
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: IVI Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2206-MAD-089-SC
Record Dates: First submitted 2024-01-11; First posted 2024-02-06 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-02

CONDITIONS: Luteinised Follicular Cyst

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group: Oral administration of letrozole (Experimental): Oral administration of letrozole 5 mg (each capsule is 2.5 mg) once a day for 5 days starting on the night of the follicular puncture. day for 5 days starting the night of the follicular puncture.
  Interventions: Drug: Administration of letrozole
- Control group: No specific treatment of letrozole (No Intervention): No specific treatment with letrozol

INTERVENTIONS:
Drug: Administration of letrozole — Oral administration of letrozole 5 mg (each capsule is 2.5 mg) once a day for 5 days starting on the night of the follicular puncture.
  Other Names: Oral administration of letrozole
  Arms: Study group: Oral administration of letrozole

SUMMARY:
The objective of this trial is to determine whether the use of letrozole during the luteal phase in oocyte donors diminishes the ovarian volume, as well as to evaluate its effect on the duration of the luteal phase, taking into account hormonal and biochemical markers.

Two groups will be established with random allocation of patients and 1:1 proportionality, as follows:

* Control group: No specific treatment.
* Study group: Oral administration of letrozole 5 mg (each capsule is 2.5 mg) once a day for 5 days starting on the night of the follicular puncture.

DETAILED DESCRIPTION:
Letrozole is a widely used drug in the context of hormone-dependent malignant tumors due to its antiestrogenic effect. Its mechanism of action allows its application to the field of Assisted Reproductive Medicine, mainly as an inductor of ovulation, by means of a blockage in the negative feedback signalization of the hypothalamus-pituitary-gonadal axis. In the last years, it has also been tested with the goals of preventing ovarian hyperstimulation syndrome (OHSS) or analyzing its effects on several endocrinological and biochemical markers such as LH, progesterone or VEGF. However, the results are inconsistent on every account. Data regarding the effect on ovarian size and the duration of the luteal phase following the administration of letrozole after the oocyte pick-up can be useful to evaluate the benefit of this drug in patients with a tendency towards hyperresponse, in which both the discomfort after the stimulation and the risk of ovarian torsion are increased.

The objective of this trial is to determine whether the use of letrozole during the luteal phase in oocyte donors diminishes the ovarian volume, as well as to evaluate its effect on the duration of the luteal phase, taking into account hormonal and biochemical markers

ELIGIBILITY:
Inclusion Criteria:

* Hyper-responsiveness to stimulation, defined as the presence of ≥18 follicles of size ≥11 mm (22-24) on the day of the last ultrasound visit prior to ovarian puncture.

Exclusion Criteria:

* Participation in another clinical study, prior to inclusion in the present study, that could affect the objectives of this study.
* Known allergy to letrozole.
* Known lactose intolerance.

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women who have been accepted into IVI's oocyte donation programme
Enrollment: 152 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
To determine ovarian volume in millilitres in oocyte donors according to whether or not they receive the treatment during the luteal phase after ovarian stimulation. | On the day of ovarian puncture, 5 days post-puncture and 10 days post-puncture.
  Difference (in millilitres) in the mean volume of the two ovaries, calculated for each ovary according to the formula for the volume of an ellipsoid

SECONDARY OUTCOMES:
To determine the levels of VEGF, VEGF/sFlt-1 ratio, LH, FSH, oestradiol, progesterone and testosterone in the plasma of oocyte donors depending on whether or not they receive the study treatment during the luteal phase. | On the day of ovarian puncture, 5 days post-puncture and 10 days post-puncture.
  To determine the difference of plasma values of VEGF, sFlt-1, oestradiol, progesterone, FSH, LH and testosterone. Ratio VEGF/sFlt-1. Continuous numerical variables.
To determine the duration of the luteal phase in oocyte donors depending on whether or not they receive the treatment under study during the luteal phase after ovarian stimulation. | On the day of ovarian puncture and 10 days post-puncture.
  To determine the difference of duration of the luteal phase, inferred by the number of days from follicular puncture to the start of the next menstrual cycle. onset of the next menstrual cycle. Discrete numerical variable.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Caballero, PhD, Principal Investigator — IVIRMA MADRID
Locations (1):
- IVI-Madrid, Madrid, Spain